CLINICAL TRIAL: NCT00714779
Title: Fluoxetine vs. Brief Psychotherapy in the Treatment of Major Depression - a Randomized Comparative Study
Brief Title: Fluoxetine vs. Brief Psychotherapy for Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: KELA (Unknown); Finnish State Grant (Unknown)
Responsible Party: Professor Hasse Karlsson, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HK123
Record Dates: First submitted 2008-07-07; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive Disorder; fluoxetine; short-term psychodynamic psychotherapy; PET
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Fluoxetine
  Interventions: Drug: Fluoxetine
- 2 (Active Comparator): Short-term psychodynamic psychotherapy
  Interventions: Behavioral: Short-term psychodynamic psychotherapy

INTERVENTIONS:
Drug: Fluoxetine — 20-40 mg / day orally
  Arms: 1
Behavioral: Short-term psychodynamic psychotherapy — 1 session / week for 16 weeks
  Arms: 2

SUMMARY:
In this study we compare two treatments for major depression - fluoxetine and brief psychodynamic psychotherapy. In addition to more traditional outcome measures, we also measure the densities of 5HT-1A and D-2 receptors before and after the treatment. The main hypothesis is that brief psychotherapy is as effective as fluoxetine.

DETAILED DESCRIPTION:
This study is a randomized comparison of two treatments for major depression - fluoxetine and brief psychodynamic psychotherapy. The patients are recruited from occupational health services and suffer from mild to moderate major depressive disorder. The treatments last for 16 weeks. The main outcome measures include HAM-D, BDI, SOFAS, Rand-36. In addition to more traditional outcome measures, we also measure the densities of 5HT-1A and D-2 receptors before and after the treatment using Positron Emission Tomography (PET) . The main hypothesis is that brief psychotherapy is as effective as fluoxetine, but differences between the treatments are seen in PET scanning.

ELIGIBILITY:
Inclusion Criteria:

* MDD (mild to moderate)
* HDRS 15 or more, age 20-60 years
* No treatment for preceding 4 months
* No DSM-IV axis I or II comorbidity
* No severe somatic illness
* No contraindications for fluoxetine treatment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2000-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
HAM-D | 0, 16 weeks, one year

CONTACTS AND LOCATIONS:
Overall Officials: Hasse Karlsson, MA, MD, PhD, Principal Investigator — University of Helsinki